CLINICAL TRIAL: NCT02496702
Title: Efficacy of Interactive Modular Tiles Training Versus "Usual Care" on Physical Attributes Among Elder Adults 70+. A Randomized Controlled Trial
Brief Title: Playware Technology for Balance Training
Acronym: IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Jari Due Jessen, PhD Student, Technical University of Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-15006703
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2017-10

CONDITIONS: Accidental Falls
Keywords: exergaming; Senior Fitness Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): The intervention is done in the form of groups of 4-5 participants per set of tiles, with 2-3 set of tiles at a time. As more set can be used it is possible to make groups of more people. The training will consist of 1.5-3 minutes of training (depending on the game) on tiles and the rest while the other 2-3 participants train (4-6 minutes of break). Then the participants will train for 1.5-3 minutes again until each participant have received a total of 13 minutes of training.
  The intervention will be done 2 times a week for 12 weeks, each session lasting 1 hour and each participant receiving 13 minutes of training each time (see training plan).
  Interventions: Device: Training on Interactive Modulare Tiles
- Control (No Intervention): No training.

INTERVENTIONS:
Device: Training on Interactive Modulare Tiles — Training with the Interactive Modulare Tiles
  Arms: Training

SUMMARY:
This study evaluates the use of Playware technology for balance training. Falling among elder is a costly problem. Research shows that training can help prevent falls. Pilot studies of the use of Interactive Modular Tiles (IMT) show that the participants can highly increase their physical abilities.

The interventions group will train using interactive modular tiles. The tiles include preprogrammed games that create playful training for the participants.

The control group will receive "usual care", which here refers to normal day activities.

The intervention will be done 2 times a week for 12 weeks, each session lasting 1 hour and each participant receiving 13 minutes of training each time.

DETAILED DESCRIPTION:
This study will investigate the use of one form of exergames called IMT how this compared to usual care of elderly people 70+. The trial will consist of two groups, one for training with the IMT and usual care that will receive the care provided to non-patients elderly, which at this moment is no additional treatment other than recommendations.

The study will be single blinded, randomized controlled trial. It will be funded by the patient@home project and Entertainment robotics. Concealed allocation and intention-to-treat analysis will be used. Measurements will be taken at baseline and after intervention. Upon acceptance the protocol will be registered in clinicaltrials.gov.

The trial's results will be reported using domains and categories described in the taxonomy developed by the Prevention of Falls Network Europe, to allow future synthesis of evidence, or study replication.

The intervention is done in the form of groups of 4-5 participants per set of tiles, with 2-3 set of tiles at a time. As more set can be used it is possible to make groups of more people. The training will consist of 1.5-3 minutes of training (depending on the game) on tiles and the rest while the other 2-3 participants train (4-6 minutes of break). Then the participants will train for 1.5-3 minutes again until each participant have received a total of 13 minutes of training.

The control group will not train.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* 70+ years

Exclusion Criteria:

* A previous diagnosis of strong dementia or a cognitive decline that prevents the understanding of simple instructions or guidelines;
* A previous stroke with a severe neurological impairment, such as loss of strength, and perceptual or language limitations;
* A severe visual deficiency;
* Inability to maintain a standing position, even with the use of a walking aid or other device;
* Participating in rehabilitative training.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University of Denmark, Kongens Lyngby, Denmark

REFERENCES:
- [Background] Lund HH, Jessen JD. Effects of Short-Term Training of Community-Dwelling Elderly with Modular Interactive Tiles. Games Health J. 2014 Oct 1;3(5):277-283. doi: 10.1089/g4h.2014.0028. PMID 25276497
- [Derived] Jessen JD, Lund HH. Study protocol: effect of playful training on functional abilities of older adults - a randomized controlled trial. BMC Geriatr. 2017 Jan 19;17(1):27. doi: 10.1186/s12877-017-0416-5. PMID 28103811

RESULTS

PARTICIPANT FLOW:
Groups:
- Training: The intervention is done in the form of groups of 4-5 participants per set of tiles, with 2-3 set of tiles at a time. As more set can be used it is possible to make groups of more people. The training will consist of 1.5-3 minutes of training (depending on the game) on tiles and the rest while the other 2-3 participants train (4-6 minutes of break). Then the participants will train for 1.5-3 minutes again until each participant have received a total of 13 minutes of training.
  The intervention will be done 2 times a week for 12 weeks, each session lasting 1 hour and each participant receiving 13 minutes of training each time (see training plan).
  Training on Interactive Modulare Tiles: Training with the Interactive Modulare Tiles
Period: Overall Study
Arm/Group | Training | Control
Started | 30 | 30
Received Allocated Intervention | 21 | 0
Did Not Receive Allocated Intervention | 9 | 0
Completed | 22 | 22
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 8 | 6
Not completed — Only partially tested | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Training | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.14 (6.69) | 82.37 (6.61) | 82.73 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 2 | 5 | 7
Timed Up and Go [Mean (Standard Deviation); unit: Seconds] | 12.24 (5.13) | 13.35 (10.10) | 12.80 (7.96)
Chair Stand [Mean (Standard Deviation); unit: Chair stands per 30 seconds] | 9.23 (4.47) | 8.77 (3.91) | 9 (4.17)
6 Minute Walking Test [Mean (Standard Deviation); unit: Meters] | 240.28 (71.21) | 237.18 (94.77) | 238.73 (83.12)
Line Walk [Mean (Standard Deviation); unit: Steps] | 2.37 (4.36) | 3.50 (2.49) | 2.93 (3.56)
Height [Mean (Full Range); unit: cm] | 1.62 [1.47 to 1.78] | 1.65 [1.49 to 1.88] | 1.63 [1.47 to 1.88]
Weight [Mean (Standard Deviation); unit: kg] | 68.33 (13.22) | 71.13 (13.34) | 69.73 (13.25)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.17 (5.21) | 26.16 (4.45) | 26.16 (4.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Test Score of 6 Minute Walking Test at Week 14.
Description: Numbers of meters that can be walked in 6 minutes around a 50-yard (45.7 meters) course. Baseline score compared to score at week 14.
Time Frame: Baseline and at week 14
Measure: Mean (95% Confidence Interval); unit: m
Arm/Group | Training | Control
Number analyzed (Participants) | 22 | 22
m | 1.07 [-13.6 to 15.7] | 0.568 [-18.2 to 19.3]

2. Primary Outcome: Change From Baseline in Test Score of 30-second Chair Stand at Week 14.
Description: Number of full stands that can be completed in 30 seconds with arms folded across chest. Baseline score compared to score at week 14.
Time Frame: Baseline and at week 14
Measure: Mean (95% Confidence Interval); unit: Full chair stands per 30 seconds
Arm/Group | Training | Control
Number analyzed (Participants) | 22 | 22
Full chair stands per 30 seconds | 2.05 [0.513 to 3.58] | 0.455 [-0.375 to 1.28]

3. Primary Outcome: Change From Baseline in Test Score of 8-Foot Up-and-Go at Week 14.
Description: Number of seconds required to get up from a seated position, walk 8 feet (2.44 meters), turn, and return to seated position. Baseline score compared to score at week 14.
Time Frame: Baseline and at week 14
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Training | Control
Number analyzed (Participants) | 22 | 22
seconds | -1.38 [-2.77 to 0.0207] | -0.0473 [-0.837 to 0.742]

4. Secondary Outcome: Change From Baseline in Test Score of Line Walk at Week 14.
Description: Number of steps a person can do on a line directly after the foot without touching outside the line. Baseline score compared to score at week 14.
Time Frame: Baseline and at week 14
Measure: Mean (95% Confidence Interval); unit: Steps
Arm/Group | Training | Control
Number analyzed (Participants) | 22 | 22
Steps | 2.23 [0.88 to 3.57] | 1.09 [-0.539 to 2.72]

5. Secondary Outcome: Change From Baseline in Test Score of Static Balance at Week 14.
Description: Static Balance will be measured using Wii Balance Board, which have proven to be a valid measure of balance (Sgró 2014). This measure will be done using an application developed by Francesco Sgró and colleagues (Sgró 2014). Baseline score compared to score at week 14.
Time Frame: Baseline and at week 14
Population: Data were not collected.
Arm/Group | Training | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Adherence to Training, Composite Outcome Measure.
Description: Adherence to the training will be measured by registering the number of times the participants participate and how much they participate at each session.
Time Frame: At week 14
Measure: Mean (95% Confidence Interval); unit: percentage of sessions
Arm/Group | Training | Control
Number analyzed (Participants) | 22 | 0
percentage of sessions | 90.6 [85.6 to 95.6] |

7. Secondary Outcome: Motivation for Training
Description: Semi-structured interviews will be done with the participant after the intervention to investigate the motivation of the IMT.
Time Frame: At week 14.
Measure: Number; unit: percentage of wanting to continue
Arm/Group | Training | Control
Number analyzed (Participants) | 20 | 0
percentage of wanting to continue | 85 |

8. Secondary Outcome: Acceptability of IMT
Description: Semi-structured interviews will be done with the participant after the intervention to investigate the acceptability of the IMT
Time Frame: At week 14.
Measure: Number; unit: percentage of happy to train on IMT
Arm/Group | Training | Control
Number analyzed (Participants) | 20 | 0
percentage of happy to train on IMT | 90 |

ADVERSE EVENTS:
Arm/Group | Training | Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes